CLINICAL TRIAL: NCT03951662
Title: Effects of Alcoholic Hepatitis on Immunological and Virological Profiles in HIV-Positive Patients
Brief Title: Immunology of HIV and Alcoholic Hepatitis
Status: Withdrawn | Type: Observational
Why Stopped: Funding ended
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Professor of Medicine, Indiana University
Other Study IDs: NIAAA 1UH2AA026218
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: HIV/AIDS; Alcoholic Hepatitis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis, Alcoholic | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC, plasma, serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With alcoholic hepatitis: HIV-positive patients receiving antiretroviral therapy and who are heavy drinkers with high bilirubin and AST levels.
  Interventions: Other: Alcoholic Hepatitis Group
- Without alcoholic hepatitis: HIV-positive patients receiving antiretroviral therapy and who are heavy drinkers without high bilirubin and AST levels.
  Interventions: Other: Heavy Drinking Controls without Hepatitis

INTERVENTIONS:
Other: Alcoholic Hepatitis Group — Alcoholic hepatitis is defined as having a total bilirubin level >3mg/dL and AST level>50U/L
  Groups: With alcoholic hepatitis
Other: Heavy Drinking Controls without Hepatitis — Normal levels of AST, ALT and total bilirubin and without evidence of cirrhosis or hepatosplenomegaly
  Groups: Without alcoholic hepatitis

SUMMARY:
This is prospective, longitudinal cohort study involving HIV-positive, antiretroviral (ART)-treated, heavy alcohol drinking participants who have and do not have alcoholic hepatitis.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the relationships between alcohol consumption and HIV-related pathogenic processes (microbial translocation, immune activation, inflammation, HIV replication, and hepatitis). Two study groups will be assembled and followed longitudinally over one year to address this objective. Group 1 will include HIV-positive, ART-treated, heavy alcohol drinkers who have alcoholic hepatitis. Group 2 will include HIV-positive, ART-treated, heavy alcohol drinkers who do not have alcoholic hepatitis. Both groups will undergo similar study procedures and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Both Groups: Age equal to or greater than 18 years
* HIV infection documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot, a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by at least one detectable HIV-1 RNA level
* Receipt of stable antiretroviral therapy of any kind for at least 90 days prior to the baseline study visit
* The most recent HIV-1 RNA level must be <200 copies/mL obtained as part of routine clinical care within 90 days prior to the main study visit
* NOTE: There is no CD4 cell count eligibility criterion for this study.
* Current alcoholism defined as >40g/day and >60g/day of alcoholic intake on average for a minimum of six months and within 90 days of the baseline visit in women and men, respectively
* For Group 1 (Alcoholic Hepatitis Group), the presence of alcoholic hepatitis is defined by

  * Per most recently obtained routine clinical care laboratories, a total bilirubin > 3mg/dL and AST >50U/L, both within 90 days of the baseline study visit
  * For Group 1, participants who have become alcohol abstinent within 14 days of the baseline visit will still be allowed to participate
* For Group 2 (Heavy drinking controls without hepatitis):

  * The most recent AST, ALT, and total bilirubin levels must be within normal limits. However, if the bilirubin level is increased due to suspected Gilbert's syndrome or due to current use of atazanavir, then the participant will be eligible.
  * There must not be evidence of current hepatosplenomegaly by examination or imaging obtained previously
  * There must not be stigmata of cirrhosis (spider angiomata, jaundice, encephalopathy, palmar erythema, ascites, intestinal varices).

Exclusion Criteria:

* Inability to complete written, informed consent
* Incarceration at the time of screening or main study visit
* Abstinence from alcohol >2 weeks prior to the baseline study visit
* Liver disease considered to be due to any etiology besides alcohol use
* Diagnosed disease or process associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosus, inflammatory bowel diseases, other collagen vascular/autoimmune diseases)
* Known active hepatitis B (defined as hepatitis B surface antigen positive with quantifiable HBV DNA viral load) or active hepatitis C (defined as quantifiable hepatitis C RNA viral load)
* Fever, defined as T ≥ 38.0C within 48 hours prior to any study visit
* Therapy for acute infection or other serious medical illnesses within 7 days of study visit
* Malignancy requiring active treatment or had completed treatment within 90 days of any study visit (excluding skin-limited Kaposi sarcoma)
* Pregnancy or breastfeeding within 14 days of any study visit
* Receipt of investigational agents, cytotoxic chemotherapy, systemic or topical glucocorticoids (of any dose), or anabolic steroids (including physiologic testosterone replacement therapy) within 14 days of study visit
* Active illicit drug use (besides marijuana) via any intake route (inhalation, smoking, injection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with HIV infection who are receiving antiretroviral therapy and who are heavy drinkers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Immune activation - Levels of sCD14, sCD163 | One year
  Levels of sCD14, sCD163

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No